CLINICAL TRIAL: NCT05215431
Title: The EFFECTS of NON-SURGICAL PERIODONTAL TREATMENT in PATIENTS with SYSTEMIC SCLEROSIS
Brief Title: Periodontal Health Status in Patients with Systemic Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Natasa Nikolic Jakoba, Clinical Professor, University of Belgrade
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unique Protocol ID: UBelgrade7
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-11

CONDITIONS: Systemic Sclerosis; Periodontitis
Keywords: systemic sclerosis; periodontitis; antioxidants; saliva
MeSH Terms: conditions — Scleroderma, Systemic; Periodontitis | interventions — Vascular Endothelial Growth Factor A; Interleukin-17; Periodontal Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- systemic sclerosis group (Experimental): Patients with established diagnoses of systemic sclerosis and periodontitis
  Interventions: Procedure: periodontal examination's, determination of salivary antioxidants and cytokine levels (VEGF, TGF-β, Il-17) in gingival crevicular fluid, Non-surgical therapy of periodontitis; Diagnostic Test: Activity of antioxidants in unstimulated saliva (GPX, SOD, UA); Diagnostic Test: Total cytokine levels (VEGF, TGF-β, Il-17) in gingival crevicular fluid; Procedure: Periodontal treatment
- periodontitis group (Experimental): Systemically healthy periodontitis patients
  Interventions: Procedure: periodontal examination's, determination of salivary antioxidants and cytokine levels (VEGF, TGF-β, Il-17) in gingival crevicular fluid, Non-surgical therapy of periodontitis; Diagnostic Test: Activity of antioxidants in unstimulated saliva (GPX, SOD, UA); Diagnostic Test: Total cytokine levels (VEGF, TGF-β, Il-17) in gingival crevicular fluid; Procedure: Periodontal treatment

INTERVENTIONS:
Procedure: periodontal examination's, determination of salivary antioxidants and cytokine levels (VEGF, TGF-β, Il-17) in gingival crevicular fluid, Non-surgical therapy of periodontitis — Periodontal parameters has been recorded on six sites of each tooth using a manual periodontal probe. Activity of antioxidants in unstimulated saliva (GPX, SOD, UA) has been determined using the colorimetric method and commercial kits. Total cytokine levels (VEGF, TGF-β, Il-17) in gingival crevicular fluid were determined using commercial ELISA (enzyme-linked immunosorbent assay) kits . The therapeutic procedure begun with ultrasonic scaling (MiniPiezon, EMS Electro Medical Systems, Switzerland), along with education and motivation of subjects to maintain oral hygiene properly. Periodontal debridement was carried out under local anesthesia, by quadrants, starting from the upper right quadrant at 7-day intervals until the completion of therapy. Instrumentation of all periodontal pockets was processed manually using specialized curettes.
Diagnostic Test: Activity of antioxidants in unstimulated saliva (GPX, SOD, UA) — Activity of antioxidants in unstimulated saliva (GPX, SOD, UA) has been determined using the colorimetric method and commercial kits.
Diagnostic Test: Total cytokine levels (VEGF, TGF-β, Il-17) in gingival crevicular fluid — Total cytokine levels (VEGF, TGF-β, Il-17) in gingival crevicular fluid were determined using commercial ELISA (enzyme-linked immunosorbent assay) kits .
Procedure: Periodontal treatment — The therapeutic procedure begun with ultrasonic scaling (MiniPiezon, EMS Electro Medical Systems, Switzerland), along with education and motivation of subjects to maintain oral hygiene properly. Periodontal debridement was carried out under local anesthesia, by quadrants, starting from the upper right quadrant at 7-day intervals until the completion of therapy. Instrumentation of all periodontal pockets was processed manually using specialized curettes.

SUMMARY:
The aim of the research will be to evaluate the effects of NSPT on clinical periodontal parameters, level of antioxidants in unstimulated saliva and the levels of biomarkers (VEGF, TGF-β, IL-17) in the GCF in SSc patients in comparison with systemically healthy controls. Twenty systemic sclerosis patients with periodontitis (SS group) and twenty systemically healthy periodontitis patients (P group) will be enrolled in the present study. The results may indicate higher periodontal destruction and antioxidant perturbations in unstimulated saliva of systemic sclerosis patients with periodontitis compared to systemically healthy periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* established diagnoses of systemic sclerosis and periodontitis (study group),
* age ≥ 18
* presence of minimum 12 teeth

Exclusion Criteria:

* concurrent inflammatory mediated rheumatic diseases
* pregnancy or lactation
* active cigarette smokers
* a history of periodontal, antibiotics or non-steroidal drug therapy in the past 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | one day
  Measuring the CAL by periodontal probe, measured in mm
Probing depth (PD) | one day
  Measuring the PD by periodontal probe, measured in mm
Gingival margin level (GML) | one day
  Measuring the GML by periodontal probe, measured in mm
The degree of gingival inflammation | one day
  The degree of gingival inflammation was assessed using the Loe and Silness (LSGI) gingival index.
plaque index (PI) | one day
  Evaluation of oral hygiene status was recorded with a Silness Loe plaque index (PI).
The concentration of vascular endothelial growth factor (VEGF) | baseline and two months after periodontal treatment
  The level of VEGF were determined using commercial ELISA (enzyme-linked immunosorbent assay) kits.
The concentration of transforming growth factor beta (TGF-β) | baseline and two months after periodontal treatment
  The level of TGF-β in gingival crevicular fluid was determined using commercial ELISA (enzyme-linked immunosorbent assay) kits at the Implant Research Center, School of Dental Medicine, University of Belgrade, following the manufacturer's instructions.
The concentration of interleukin (IL)-17 | baseline and two months after periodontal treatment
  interleukin (IL)-17 was determined using commercial ELISA (enzyme-linked immunosorbent assay) kits at the Implant Research Center, School of Dental Medicine, University of Belgrade, following the manufacturer's instructions.
The concentration of glutathion peroxidase (GPX) | one day
  Activity level of GPX, determined using the colorimetric method and commercial kits.
The concentration of uric acid (UA) | one day
  Activity level of UA, determined using the colorimetric method and commercial kits.
The concentration of superoxide dismutase (SOD) | one day
  Activity level of SOD, determined using the colorimetric method and commercial kits.
The concentration of tumor necrosis factor alpha | baseline and two months after periodontal treatment
The concentration of C reactive protein | baseline and two months after periodontal treatment
Erythrocyte sedimentation rate (ESR) | baseline and two months after periodontal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Natasa Nikolic Jakoba, DDS, PhD, Principal Investigator — School of Dental Medicine, University of Belgrade, Serbia
Locations (1):
- Department of Periodontology and Oral medicine, School of Dental Medicine, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No